CLINICAL TRIAL: NCT00836342
Title: Comparison of Skin Carotenoid Levels Between Subjects With History of Cutaneous Squamous Cell Carcinoma and Subjects With History of Basal Cell Carcinoma Versus a Control Group
Brief Title: Correlation Between Skin Carotenoid Levels and Previous History of Skin Cancer
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Nu Skin Enterprises (Industry)
Responsible Party: Principal Investigator, Alexandra Kimball, Director, Clinical Unit for Research Trials in Skin, Massachusetts General Hospital
Other Study IDs: 2008-P-002240
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-06

CONDITIONS: Skin Cancer; Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: Non-melanoma skin cancer; Basal cell carcinoma; Squamous cell carcinoma
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Previous history of SCC: Participants had previous history of SCC
- Previous history of BCC: Participants had previous history of BCC
- Control: Participants had no previous history of squamous cell carcinoma or basal cell carcinoma

SUMMARY:
The purpose of this study is to determine the difference of skin carotenoid levels between subjects with previous squamous cell carcinomas (SCC), subjects with previous basal cell carcinomas (BCC) and a control group.

DETAILED DESCRIPTION:
There has been experimental and clinical research evaluating association of different carotenoids and incidence of malignancies, including Non- Melanoma Skin Cancer (NMSC). An easy and inexpensive way to determine which subjects would benefit from supplementation with carotenoids or retinoids could be the measurement of skin carotenoid levels.The least invasive way to perform it is through Raman spectroscopy which is a technique that uses a laser light that can be used to quantify carotenoids on the skin. We will compare the skin carotenoid levels of subjects with previous history of SCC or BCC and subjects without history of previous NMSC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 50 and 75 years old without history of previous SCC or BCC.
* Fitzpatrick skin types I-IV.
* Willing and able to understand and sign informed consent.
* Able to complete study and comply with study procedures

Exclusion Criteria:

* Regular ingestion of supplements containing carotenoids or vitamin A in the past 4 weeks.
* Use of topical retinoids in the past 4 weeks.
* Treatment with systemic retinoids in the past 6 months.
* Dermatologic conditions that require the use of interfering topical or systemic therapy or that might interfere with study assessments such as, but not limited to, palmar psoriasis, hand dermatitis or palmo-plantar keratoderma.
* Previous history of psoriasis.
* Clinically significant abnormal findings or conditions, which might, in the opinion of the Principal Investigator, interfere with study evaluations or pose a risk to subject safety during the study.
* Subjects who are known to be pregnant or planning a pregnancy.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research population were recruited from Massachusetts General Hospital dermatology clinics.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B Kimball, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Clinical Unit for Research Trials in Skin - MGH, Boston, Massachusetts, United States

REFERENCES:
- [Background] Bath-Hextall F, Leonardi-Bee J, Somchand N, Webster A, Delitt J, Perkins W. Interventions for preventing non-melanoma skin cancers in high-risk groups. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD005414. doi: 10.1002/14651858.CD005414.pub2. PMID 17943854
- [Background] Santamaria L, Bianchi A. Cancer chemoprevention by supplemental carotenoids in animals and humans. Prev Med. 1989 Sep;18(5):603-23. doi: 10.1016/0091-7435(89)90033-9. PMID 2694158
- [Background] Heinen MM, Hughes MC, Ibiebele TI, Marks GC, Green AC, van der Pols JC. Intake of antioxidant nutrients and the risk of skin cancer. Eur J Cancer. 2007 Dec;43(18):2707-16. doi: 10.1016/j.ejca.2007.09.005. Epub 2007 Nov 7. PMID 17988857
- [Background] Frieling UM, Schaumberg DA, Kupper TS, Muntwyler J, Hennekens CH. A randomized, 12-year primary-prevention trial of beta carotene supplementation for nonmelanoma skin cancer in the physician's health study. Arch Dermatol. 2000 Feb;136(2):179-84. doi: 10.1001/archderm.136.2.179. PMID 10677093
- [Background] Ermakov IV, Ermakova MR, McClane RW, Gellermann W. Resonance Raman detection of carotenoid antioxidants in living human tissues. Opt Lett. 2001 Aug 1;26(15):1179-81. doi: 10.1364/ol.26.001179. PMID 18049555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from May 2009 to December 2011. Subjects were recruited from dermatology medical and surgery clinics at the Massachusetts General Hospital.
Pre-assignment Details: Patients were enrolled in the study if they had a history of cutaneous basal cell carcinoma or cutaneous squamous cell carcinoma but were excluded if they had a history of both basal cell carcinoma and squamous cell carcinoma. Participants were also excluded if they were using retinoids or taking a multivitamin regularly for less than 5 yrs.
Groups:
- Previous History of SCC: Participants had previous history of squamous cell carcinoma
- Previous History of BCC: Participants had previous history of basal cell carcinoma
- Control Group: Participants had no history of squamous cell carcinoma or basal cell carcinoma
Period: Overall Study
Arm/Group | Previous History of SCC | Previous History of BCC | Control Group
Started | 22 | 23 | 36
Completed | 22 | 23 | 36
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Previous History of SCC | Previous History of BCC | Control Group | Total
Number analyzed (Participants) | 22 | 23 | 36 | 81
Age Continuous [Mean (Full Range); unit: years]
  Mean age | 63.9 [50 to 75] | 60.9 [50 to 75] | 57.4 [50 to 75] | 60.2 [50 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 30 | 55
  Male | 10 | 10 | 6 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 22 | 23 | 31 | 76
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Skin Carotenoid Levels in Subjects With History of Squamous Cell Carcinoma Versus Control Subjects
Description: Mean carotenoid levels in subjects with a history of squamous cell carcinoma were compared to mean carotenoid levels in control subjects without a history of nonmelanoma skin cancer.
Time Frame: baseline
Population: Participants that passed inclusion criteria and consented for skin carotenoid measurement were analyzed.
Measure: Mean (Standard Deviation); unit: Raman spectroscopy intensity counts
Groups:
- Control Group: Participants had no previous history or squamous cell carcinoma or basal cell carcinoma
Arm/Group | Previous History of SCC | Control Group
Number analyzed (Participants) | 22 | 36
Raman spectroscopy intensity counts | 27,635 (12,013) | 31,219 (13,320)
Statistical Analysis 1: Comparison: Previous History of SCC vs Control Group; Null hypothesis: There is no difference in mean carotenoid levels between subjects with a history of squamous cell carcinom and control subjects; Test type: Superiority or Other; p = 0.31, t-test, 2 sided

2. Secondary Outcome: Skin Carotenoid Levels in Subjects With History of Squamous Cell Carcinoma Versus Subjects With History of Basal Cell Carcinoma
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Raman spectroscopy intensity counts
Arm/Group | Previous History of SCC | Previous History of BCC
Number analyzed (Participants) | 22 | 23
Raman spectroscopy intensity counts | 27,635 (12,013) | 25,031 (12,825)
Statistical Analysis 1: Comparison: Previous History of SCC vs Previous History of BCC; Test type: Superiority or Other; p = 0.49, t-test, 2 sided

3. Secondary Outcome: Skin Carotenoid Levels in Subjects With History of Basal Cell Carcinoma Versus Control Group
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Raman spectrocopy intensity counts
Groups:
- Control Group: Participants had no history of previous squamous cell carcinoma or basal cell carcinoma
Arm/Group | Previous History of BCC | Control Group
Number analyzed (Participants) | 23 | 36
Raman spectrocopy intensity counts | 25,031 (12,825) | 31,219 (13,320)
Statistical Analysis 1: Comparison: Previous History of BCC vs Control Group; Test type: Superiority or Other; p = 0.09, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Previous History of SCC | Previous History of BCC | Control Group
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/36
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/36

LIMITATIONS AND CAVEATS:
Limitations include a small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No